CLINICAL TRIAL: NCT02027545
Title: Promoting Veteran-Centered Colorectal Cancer Screening
Acronym: PROM-IS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other); Memorial Sloan Kettering Cancer Center (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 12-411
Record Dates: First submitted 2013-12-18; First posted 2014-01-06 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer
Keywords: cancer screening; decision making
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: A cluster-randomized (by provider) pragmatic trial of the patient-centered intervention versus pragmatic control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decision Aid (Experimental): Patients of primary care providers randomly assigned to the Decision Aid intervention (DA) that includes an individualized decision aid, provider education, and modified performance measure/reminder.
  Interventions: Behavioral: Decision Aid; Behavioral: Provider Education; Behavioral: Performance Measure Modification
- No Decision Aid (Other): Patients of primary care providers will be randomly assigned to the pragmatic control (PC) that includes provider education and modified performance measure/reminder, but no decision aid.
  Interventions: Behavioral: Provider Education; Behavioral: Performance Measure Modification; Behavioral: Simple Informational Booklet

INTERVENTIONS:
Behavioral: Decision Aid — Printed booklet comprising educational information about benefits and harms of screening, individualized estimates of benefits and harms of screening, and values clarification exercise
  Arms: Decision Aid
Behavioral: Provider Education — Providers of patients in both arms of the study will be given an educational module about recent data on the benefits and harms of screening how these data fit in with existing population-centered guidelines.
Behavioral: Performance Measure Modification — The clinical reminder system will be modified so to facilitate documentation of informed decision making about CRC screening, including specific reasons for not screening. Additionally, providers who indicate a specific exception for not screening (using the modified clinical reminder) will be considered as satisfying the requirements and will not be penalized in terms of performance pay, and will be removed from feedback reports that encourage population screening.
Behavioral: Simple Informational Booklet — A simple informational booklet explaining colorectal cancer screening and current screening recommendations.
  Arms: No Decision Aid

SUMMARY:
Systematic efforts to improve colorectal cancer screening use in the VA Healthcare System have resulted in an increase in not only appropriate, but also inappropriate use of screening. The purpose of this study is to test a new, more patient-centered approach to colon cancer screening. In older individuals (ages 70 to 75) who are "due" for screening, the investigators will provide education on the benefits and harms of colon cancer screening. But instead of simply providing these patients with "average" information about these benefits, the investigators will give them information that takes into account their personal characteristics (e.g., age, gender), overall health, and screening history and therefore applies to them more personally. The investigators will also work with the health system to create time and space for patient and doctor to discuss whether screening is the right choice for each individual. This way, patients can make an informed choice about what is right for them, with the help of their doctor. In the future, the results of this study will help patients make more informed screening decisions, especially when the benefits of screening may be uncertain for them personally.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) screening is a widely recommended, evidence-based preventive service that has traditionally been underused. Over the last decade, organized efforts by the Veterans Health Administration (VHA) to increase population screening among Veterans have been successful. But these population-centered efforts have increased screening utilization in a way that is not always concordant with screening benefit, particularly among older Veterans, those with comorbid illness, and those who have previously been screened. As patients get older, acquire health problems, and undergo negative screening tests, the benefit of screening decreases and the potential harm of screening increases. Yet, existing population-centered efforts fail to adequately inform these patients about this changing balance in benefit and harm, often yielding screening utilization that is discordant with benefit. The purpose of this study is to test a more Veteran-centered approach to screening in these individuals, one that encourages informed, personalized screening decisions based on individual values, preferences, and health status.

The 3-part intervention consists of: (1) a decision aid to help Veterans make informed screening decisions; (2) education for providers on how the benefits of screening vary between patients; and (3) modification of clinical reminder systems to allow Veterans to make informed decisions about screening. The intervention will be tested in a pragmatic cluster-randomized controlled trial (cluster = provider) at two sites in the VA Ann Arbor Healthcare System. The primary outcome will be whether screening was ordered at the clinic visit. The investigators will also assess the appropriateness of screening orders (i.e., whether screening is ordered in concordance with screening benefit), conceptual understanding of screening, elements of informed decision-making addressed in the screening discussion, and screening utilization at 6 months.

Note: In March 2023, during preparation of the final manuscript for submission for publication, the study team noted that one subject in the intervention arm had undergone colorectal cancer screening immediately prior to the study visit (but after assessment for study eligibility), making the subject ineligible (protocol violation). Study results were re-analyzed accordingly and updated on clinicaltrials.gov (analyzed N=431 rather than N=432). Additionally, a data entry error was noted on clinicaltrials.gov for the secondary outcome of screening utilization (control N=96 rather than control N=95).

ELIGIBILITY:
Inclusion Criteria:

* Aged 70-75 years
* Due for screening according to the 2008 USPSTF colorectal cancer screening guideline
* Scheduled for a non-urgent primary care visit at the Ann Arbor VA Medical Center or Toledo VA Community-Based Outpatient Clinic

Exclusion Criteria:

* Increased risk for colorectal cancer (and therefore not candidates for average-risk screening)
* Limited life expectancy (e.g., enrolled in hospice or diagnosed with metastatic cancer), or for whom the provider previously documented an intention not to pursue screening.
* Scheduled for an appointment where stimulating a discussion about screening is likely to be inappropriate: urgent appointment (for acute complaints), follow-up visit after hospitalization
* Have a condition that would impair his/her ability to participate in the study: dementia or other cognitive impairment, visual impairment, non-English speaking
* Assigned to an ineligible primary care provider (i.e., the provider did not consent to the study)
* Have Medical Guardian who makes decisions for the patient about his/her care

Ages: 70 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 436 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sameer D. Saini, MD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saini SD, van Hees F, Vijan S. Smarter screening for cancer: possibilities and challenges of personalization. JAMA. 2014 Dec 3;312(21):2211-2. doi: 10.1001/jama.2014.13933. No abstract available. PMID 25461993
- [Result] van Hees F, Saini SD, Lansdorp-Vogelaar I, Vijan S, Meester RG, de Koning HJ, Zauber AG, van Ballegooijen M. Personalizing colonoscopy screening for elderly individuals based on screening history, cancer risk, and comorbidity status could increase cost effectiveness. Gastroenterology. 2015 Nov;149(6):1425-37. doi: 10.1053/j.gastro.2015.07.042. Epub 2015 Aug 4. PMID 26253304
- [Result] Caverly TJ, Kerr EA, Saini SD. Delivering Patient-Centered Cancer Screening: Easier Said Than Done. Am J Prev Med. 2016 Jan;50(1):118-121. doi: 10.1016/j.amepre.2015.08.003. Epub 2015 Oct 9. No abstract available. PMID 26456874
- [Result] Veenstra CM, Abrahamse P, Wagner TH, Hawley ST, Banerjee M, Morris AM. Employment benefits and job retention: evidence among patients with colorectal cancer. Cancer Med. 2018 Mar;7(3):736-745. doi: 10.1002/cam4.1371. Epub 2018 Feb 23. PMID 29473344
- [Derived] Saini SD, Lewis CL, Kerr EA, Zikmund-Fisher BJ, Hawley ST, Forman JH, Zauber AG, Lansdorp-Vogelaar I, van Hees F, Saffar D, Myers A, Gauntlett LE, Lipson R, Kim HM, Vijan S. Personalized Multilevel Intervention for Improving Appropriate Use of Colorectal Cancer Screening in Older Adults: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2023 Dec 1;183(12):1334-1342. doi: 10.1001/jamainternmed.2023.5656. PMID 37902744
- See also: Click here for more information about this study: Promoting Veteran-Centered Colorectal Cancer Screening — http://www.screeningdecision.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Decision Aid: Patients of primary care providers randomly assigned to the intervention which included 1) a decision aid; 2) modified performance measure/reminder; and, 3) provider education.
  1. A printed booklet comprising educational information about benefits and harms of screening, individualized estimates of benefits and harms of screening, and a values clarification exercise.
  2. The clinical reminder system was modified to facilitate documentation of informed decision making about CRC screening, including specific reasons for not screening. Providers who indicated an exception for not screening a patient were considered as satisfying the requirements and were not penalized in terms of performance pay. Additionally, the patient was removed from provider feedback reports that encourage population screening.
  3. Providers were given information about recent data on the benefits and harms of screening & how these data fit in with existing population-centered guidelines.
- No Decision Aid: Patients of primary care providers randomly assigned to the pragmatic control which included 1) a simple booklet in place of the decision aid; 2) modified performance measure/reminder; and, 3)provider education.
  1. A simple informational booklet explaining colorectal cancer (CRC) screening and current screening recommendations.
  2. The clinical reminder system was modified to facilitate documentation of informed decision making about CRC screening, including specific reasons for not screening. Providers who indicated a specific exception for not screening a patient were considered as satisfying the requirements and were not penalized in terms of performance pay. Additionally, the patient was removed from provider feedback reports that encourage population screening.
  3. Providers were given information about recent data on the benefits and harms of screening & how these data fit in with existing population-centered guidelines.
Period: Overall Study
Arm/Group | Decision Aid | No Decision Aid
Started | 261 | 175
Completed | 258 | 173
Not Completed | 3 | 2
Not completed — Failed to sign HIPAA | 0 | 2
Not completed — Failed to attend study visit | 2 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Decision Aid: Patients of primary care providers randomly assigned to the pragmatic control which included 1) a simple booklet in place of the decision aid; 2) modified performance measure/reminder; and, 3) provider education.
  1. A simple informational booklet explaining colorectal cancer (CRC) screening and current screening recommendations.
  2. The clinical reminder system was modified to facilitate documentation of informed decision making about CRC screening, including specific reasons for not screening. Providers who indicated a specific exception for not screening a patient were considered as satisfying the requirements and were not penalized in terms of performance pay. Additionally, the patient was removed from provider feedback reports that encourage population screening.
  3. Providers were given information about recent data on the benefits and harms of screening & how these data fit in with existing population-centered guidelines.
- Total: Total of all reporting groups
Arm/Group | Decision Aid | No Decision Aid | Total
Number analyzed (Participants) | 258 | 173 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] — Defined as age at date of study visit. Date of birth electronically collected from administrative health record data.
  years | 71.5 (1.6) | 71.7 (1.7) | 71.5 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Data were collected from electronic administrative health record information.
  Participants
    Female | 5 | 2 | 7
    Male | 253 | 171 | 424
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Self-reported race via survey.
  Participants
    White | 226 | 148 | 374
    Black or African American | 18 | 8 | 26
    Native Hawaiian or other Pacific Islander | 0 | 1 | 1
    Native Indian or Alaskan Native | 3 | 2 | 5
    Missing | 11 | 14 | 25
Region of Enrollment [Count of Participants; unit: Participants] — Mailing address was collected via electronic administrative health record data.
  Participants
    United States | 258 | 173 | 431
Prior Screening [Count of Participants; unit: Participants] — Data were collected from electronic administrative health record information.
  Participants
    None | 50 | 30 | 80
    FOBT/FIT | 165 | 111 | 276
    Colonoscopy | 43 | 32 | 75
Screening Benefit [Count of Participants; unit: Participants] — Categorized distribution of screening benefit. Screening benefit is defined as colorectal cancers prevented per 1,000 patients screened.
  To create this subject-specific measure, we used a previously published simulation model to estimate the benefit of screening for individual patients according to age, prior screening, sex, and comorbidity.
  Participants
    Participants with Screening Benefit 0-4.9 | 69 | 38 | 107
    Participants with Screening Benefit 5-9.9 | 86 | 67 | 153
    Participants with Screening Benefit 10-14.9 | 57 | 40 | 97
    Participants with Screening Benefit 15-19.9 | 7 | 2 | 9
    Participants with Screening Benefit 20-24.9 | 8 | 4 | 12
    Participants with Screening Benefit 25-29.9 | 11 | 9 | 20
    Participants with Screening Benefit 30-35.0 | 20 | 13 | 33
Mean Benefit from Screening [Mean (Standard Deviation); unit: Cancers prevented per 1,000 pts screened] — Mean screening benefit is defined as colorectal cancers prevented per 1,000 patients screened.
  To create this subject-specific measure, we used a previously published simulation model to estimate the benefit of screening for individual patients according to age, prior screening, sex, and comorbidity.
  Cancers prevented per 1,000 pts screened | 11.3 (8.1) | 11.3 (8.0) | 11.3 (8.1)
Marital Status [Count of Participants; unit: Participants] — Current marital status; self-report via survey
  Participants
    Married | 162 | 108 | 270
    Separated/Divorced | 54 | 37 | 91
    Never Married | 17 | 4 | 21
    Widowed | 17 | 15 | 32
    Missing | 8 | 9 | 17
Education [Count of Participants; unit: Participants] — Highest level of education obtained; self-report via survey
  Participants
    Did not complete high school | 13 | 8 | 21
    High school/GED | 80 | 44 | 124
    Vocational, technical, or business training | 28 | 25 | 53
    1-3 years of college | 80 | 47 | 127
    Graduated college or 4 or more years of college | 32 | 23 | 55
    Graduate or professional school | 16 | 18 | 34
    Missing | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With CRC Screening Ordered
Description: The primary dependent variable in the analysis was whether screening was ordered within two weeks after the clinic visit (dichotomous). Screening orders were determined by manual record review of electronic health records.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid | No Decision Aid
Number analyzed (Participants) | 258 | 173
Participants | 162 | 114
Statistical Analysis 1: Comparison: Decision Aid vs No Decision Aid; Test type: Superiority; p = 0.491, Regression, Logistic

2. Secondary Outcome: Concordance Between Screening Orders and Screening Benefit
Description: Defined as the degree to which screening orders align with expected screening benefit, such that individuals with low screening benefit receive screening orders at a lower rate than those with high screening benefit.
  We hypothesized that Veterans randomized to the intervention (decision aid) would receive screening orders that were more concordant with screening benefit than those randomized to the control. The expected benefit of screening (reduction in CRC incidence) was calculated using the MISCAN-Colon model. For a given patient, this value was a function of age, gender, health status, and prior screening history. The regression analysis included screening orders as the dependent variable, and, study arm, expected benefit, and an interaction term between study arm and expected benefit as the independent variables. The p-value reported is for the interaction term.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid | No Decision Aid
Number analyzed (Participants) | 258 | 173
Participants | 162 | 114
Statistical Analysis 1: Comparison: Decision Aid vs No Decision Aid; Test type: Superiority; p = 0.049, Regression, Logistic

3. Secondary Outcome: Number of Participants With CRC Screening Utilized
Description: Screening test completion was collected through manual review of electronic medical records.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid | No Decision Aid
Number analyzed (Participants) | 256 | 173
Participants | 106 | 96

ADVERSE EVENTS:
Time Frame: Serious and other (not including serious) adverse events were not collected/assessed as part of this electronic health record review and survey study.
Description: There was no contact with subjects for the electronic health record review component of the study, thus, adverse event information was not collected. The survey component examined patient reactions to educational materials and their recent primary care provider visit; adverse event data was not collected.
Arm/Group | Decision Aid | No Decision Aid
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Veteran population, low numbers of women and underrepresented minorities

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/45/NCT02027545/Prot_SAP_000.pdf